CLINICAL TRIAL: NCT03450629
Title: A Randomized, Multi-Center, Investigator-Masked, Parallel Group, Equivalence Study of Once Daily Brimonidine Tartrate Ophthalmic Suspension Compared With Three Times Daily ALPHAGAN-P® in Subjects With Open Angle Glaucoma, or Ocular Hypertension
Brief Title: Evaluation of Safety and Efficacy of PDP-716
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLR_16_33
Record Dates: First submitted 2018-02-21; First posted 2018-03-01 (Actual); Results first posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PDP-716 (Experimental)
  Interventions: Drug: Brimonidine Tartrate Ophthalmic Suspension
- Brimonidine Tartrate Ophthalmic Solution (Active Comparator)
  Interventions: Drug: Brimonidine Tartrate Ophthalmic Solution

INTERVENTIONS:
Drug: Brimonidine Tartrate Ophthalmic Suspension — PDP-716
  Arms: PDP-716
Drug: Brimonidine Tartrate Ophthalmic Solution — Three Times Brimonidine Tartrate Ophthalmic Solution
  Arms: Brimonidine Tartrate Ophthalmic Solution

SUMMARY:
The study will be conducted to evaluate the efficacy and safety of topical administration of PDP-716 compared with brimonidine tartrate ophthalmic solution.

ELIGIBILITY:
Inclusion Criteria:

1. Be male or female, of 2 years of age or older
2. Have open-angle glaucoma or ocular hypertension in both the eyes
3. Be able and willing to follow study instructions and complete all required visits.

Exclusion Criteria:

1. Females who are pregnant/lactating.
2. Have uncontrolled systemic disease which might interfere with the study
3. Any known allergy or sensitivity to the study medications or their components
4. Any other clinically relevant abnormality

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (47):
- United States (47):
  - SPARC Site 4, Chandler, Arizona
  - SPARC Site 5, Prescott, Arizona
  - SPARC Site 3, Sun City, Arizona
  - SPARC Site 38, Burbank, California
  - SPARC Site 44, Glendale, California
  - SPARC Site 45, Glendale, California
  - SPARC Site 43, Mission Hills, California
  - SPARC Site 1, Newport Beach, California
  - SPARC Site 14, Santa Barbara, California
  - SPARC Site 47, Torrance, California
  - SPARC Site 7, Colorado Springs, Colorado
  - SPARC Site 11, Coral Springs, Florida
  - SPARC Site 29, Deerfield Beach, Florida
  - SPARC Site 34, Fort Myers, Florida
  - SPARC Site 46, Hollywood, Florida
  - SPARC Site 21, Jacksonville, Florida
  - SPARC Site 35, Miami, Florida
  - SPARC Site 27, Miami, Florida
  - SPARC Site 10, Miami, Florida
  - SPARC Site 16, Miami, Florida
  - SPARC Site 19, Miami, Florida
  - SPARC Site 25, Miami, Florida
  - SPARC Site 41, Pompano Beach, Florida
  - SPARC Site 18, Tampa, Florida
  - SPARC Site 42, Atlanta, Georgia
  - SPARC Site 2, Morrow, Georgia
  - SPARC Site 22, Roswell, Georgia
  - SPARC Site 12, Chicago, Illinois
  - SPARC Site 23, Paducah, Kentucky
  - SPARC Site 40, Bowie, Maryland
  - SPARC Site 28, Kansas City, Missouri
  - SPARC Site 48, Kansas City, Missouri
  - SPARC Site 31, St Louis, Missouri
  - SPARC Site 15, Poughkeepsie, New York
  - SPARC Site 36, Rochester, New York
  - SPARC Site 30, Gastonia, North Carolina
  - SPARC Site 9, High Point, North Carolina
  - SPARC Site 17, Winston-Salem, North Carolina
  - SPARC Site 33, Fargo, North Dakota
  - SPARC Site 37, Cincinnati, Ohio
  - SPARC Site 8, Cleveland, Ohio
  - SPARC Site 24, Cranberry Township, Pennsylvania
  - SPARC Site 32, Memphis, Tennessee
  - SPARC Site 39, Houston, Texas
  - SPARC Site 13, Mission, Texas
  - SPARC Site 20, San Antonio, Texas
  - SPARC Site 26, Saint Albans, Vermont

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PDP-716: Brimonidine tartrate 0.35% ophthalmic suspension (SPARC), QD
- Brimonidine Tartrate Ophthalmic Solution: Brimonidine tartrate 0.1% ophthalmic solution (Alphagan P® 0.1%), TID
Period: Overall Study
Arm/Group | PDP-716 | Brimonidine Tartrate Ophthalmic Solution
Started | 341 | 341
Completed (Completed Visit 5) | 293 | 307
Not Completed | 48 | 34
Not completed — Adverse Event | 15 | 14
Not completed — Physician Decision | 2 | 2
Not completed — Lack of Efficacy | 2 | 0
Not completed — Lost to Follow-up | 4 | 2
Not completed — No Longer Meets Eligibility Criteria | 0 | 1
Not completed — Non-Compliance With Study Drug | 2 | 1
Not completed — Protocol Violation | 11 | 8
Not completed — Withdrawal by Subject | 12 | 6

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- PDP-716: Brimonidine Tartrate Ophthalmic Suspension
- Total: Total of all reporting groups
Arm/Group | PDP-716 | Brimonidine Tartrate Ophthalmic Solution | Total
Number analyzed (Participants) | 337 | 341 | 678
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (10.70) | 66.4 (10.96) | 66.3 (10.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199 | 200 | 399
  Male | 138 | 141 | 279
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 55 | 107
  Not Hispanic or Latino | 283 | 285 | 568
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 0 | 4
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 167 | 159 | 326
  White | 162 | 178 | 340
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Intraocular Pressure
Time Frame: Week 12 8 AM, 10 AM and 4 PM
Population: Per-Protocol Population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | PDP-716 | Brimonidine Tartrate Ophthalmic Solution
Number analyzed (Participants) | 258 | 265
mmHg
  8 AM +/- 30 min | 20.35 (3.746) | 20.79 (3.724)
  10 AM +/- 30 min | 17.38 (3.401) | 18.31 (18.31)
  4 PM +/- 30 min | 17.99 (3.309) | 17.57 (3.579)
Statistical Analysis 1: Comparison: PDP-716 vs Brimonidine Tartrate Ophthalmic Solution; Test type: Equivalence — 8 AM +/- 30 min; p = 0.0006, t-test, 2 sided
Statistical Analysis 2: Comparison: PDP-716 vs Brimonidine Tartrate Ophthalmic Solution; Test type: Equivalence — 10 AM +/- 30 min; p = 0.0291, t-test, 2 sided
Statistical Analysis 3: Comparison: PDP-716 vs Brimonidine Tartrate Ophthalmic Solution; Test type: Equivalence — 4 PM +/- 30 min; p = 0.0002, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | PDP-716 | Brimonidine Tartrate Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/337 | 0/341
Serious Adverse Events (participants affected / at risk) | 1/337 | 3/341
Other Adverse Events (participants affected / at risk) | 63/337 | 38/341
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PDP-716 (N=337) | Brimonidine Tartrate Ophthalmic Solution (N=341)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Large cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PDP-716 (N=337) | Brimonidine Tartrate Ophthalmic Solution (N=341)
Somnolence (Nervous system disorders) | 32 (32) | 21 (21)
Conjunctival hyperaemia (Eye disorders) | 8 (8) | 6 (6)
Conjunctivitis (Infections and infestations) | 15 (15) | 11 (11)
Vision blurred (Eye disorders) | 9 (9) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-09-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT03450629/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-22): https://cdn.clinicaltrials.gov/large-docs/29/NCT03450629/SAP_001.pdf